CLINICAL TRIAL: NCT01939795
Title: Effect of Physical Training Combined Cardiac Resynchronization Therapy in Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Thaís Simões Nobre Pires Santos, Phd student, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PT & CRT
Record Dates: First submitted 2013-03-27; First posted 2013-09-11 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Heart Failure
Keywords: cardiac resynchronization therapy (CRT)
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy People (No Intervention): Control group
- Untrained CRT (Experimental): Untrained CRT patients
  Interventions: Other: exercise training and/or CRT
- Exercise trained + CRT (Experimental): Exercise-trained CRT patients
  Interventions: Other: exercise training and/or CRT

INTERVENTIONS:
Other: exercise training and/or CRT — Three 40-minute exercise sessions per week on a treadmill for four months
  Other Names: Untrained CRT patients; Exercise-trained CRT patients
  Arms: Exercise trained + CRT; Untrained CRT

SUMMARY:
The investigators hypothesis that exercise training would potentiate the effects of cardiac resynchronization therapy in heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* QRS> 150 ms or 120-150ms associated dyssynchrony
* The etiology can be idiopathic, ischemic, hypertensive and Chagas' disease
* Ejection fraction <35%
* The optimal pharmacological treatment for heart failureExclusion Criteria:

Exclusion Criteria:

* Patients with pulmonary diseases, neurological diseases, renal, skeletal muscle diseases
* Patients with contraindications to implant a cardiac pacemaker
* Pregnancy
* New York Heart Association functional class IV
* Atrial fibrillation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Sympathetic nerve activity | 4 months
  Sympathetic nerve activity will be assessed by microneurography

SECONDARY OUTCOMES:
Peak oxygen consumption | 4 months
  Peak oxygen consumption will be determined by cardiopulmonary exercise testing
Quality of life | 4 months
  Quality of life will be assessed by questionnaire
Blood inflammatory markers | 4 months
  Blood inflammatory markers will be assessed by venipuncture
skeletal muscle strength | 4 months
  Muscular evaluation will be done muscle gene expression
Muscle Blood Flow | 4 months
  Forearm blood flow will be assessed by venous occlusion plethysmography

CONTACTS AND LOCATIONS:
Overall Officials: Carlos E Negrao, Phd, Principal Investigator — InCor, HCFMUSP
Locations (1):
- Thais Simoes Nobre Pires Santos, São Paulo, São Paulo, Brazil